CLINICAL TRIAL: NCT05763472
Title: Molecular Landscape Involved in the Onset of Breast Cancer in Patients With Germline BRCA-1/2 Mutations, During or After Therapy With Platinum-based Agents and/or PARP-inhibitors for Ovarian Cancer
Brief Title: Breast Cancer After Ovarian Cancer During and/or After Therapy: Genomic Evaluation
Acronym: Gen-eva
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Fondazione Policlinico Universitario Agostino Gemelli IRCCS (Other)
Responsible Party: Sponsor
Other Study IDs: 4817
Record Dates: First submitted 2023-02-28; First posted 2023-03-10 (Actual); Last update posted 2023-03-10 (Actual); Status verified 2023-02

CONDITIONS: BRCA-Associated Breast Carcinoma
Keywords: BRCA1/2; Breast cancer; Ovarian cancer; Platinum salts; PARP inhibitors
MeSH Terms: conditions — Breast Neoplasms; Ovarian Neoplasms | interventions — High-Throughput Nucleotide Sequencing

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients with germline BRCA1/2 patitents: Women with germline BRCA-1/2 mutations, previously treated or undergoing treatment with platinum-based chemotherapy and/or PARP inhibitors for ovarian cancer, who have developed breast cancer, subjected to genomic profiling of breast and ovarian tumor samples.
  Interventions: Genetic: Next-generation sequencing (NGS) assay TruSight Oncology 500 (TSO 500).

INTERVENTIONS:
Genetic: Next-generation sequencing (NGS) assay TruSight Oncology 500 (TSO 500). — Next-generation sequencing (NGS) analysis with TruSight Oncology 500 (TSO 500) is performed on tumor samples from breast and ovarian cancer of the enrolled patients.

SUMMARY:
This study will investigate, in patients with germline BRCA-1/2 mutations and breast cancer, arising during and / or after treatment with platinum-based chemotherapy and / or with PARP-inhibitors for ovarian cancer, the presence of molecular alterations potentially involved in the mechanisms of resistance to antineoplastic treatment on breast and ovarian tumor tissue.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent.
* Age older than 18 years.
* Germline BRCA1/2 mutation.
* Histologically confirmed ovarian cancer treated with platinum-based chemotherapy and/or PARP inhibitors.
* Histologically confirmed breast cancer occurred during or after therapy with platinum-based agents and/or PARP-inhibitors for ovarian cancer.
* Availability of FFPE breast and ovarian tumor samples.

Exclusion Criteria:

* Other malignancies in the last 2 years.
* Prior chemotherapy or radiation therapy for other malignancies.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with germline BRCA-1/2 mutations and breast cancer, arising during and / or after treatment with platinum-based chemotherapy and / or with PARP-inhibitors for ovarian cancer
Sampling Method: Non-Probability Sample
Enrollment: 10 (Estimated)
Dates: Start 2022-03-01 (Actual); Primary Completion 2023-06-01 (Estimated); Study Completion 2023-06-01 (Estimated)

PRIMARY OUTCOMES:
Breast somatic mutations | 15 months
  To describe the presence of somatic mutations on breast tumor tissue, in patients with breast cancer arising during or after treatment with platinum-based chemotherapy or PARP-inhibitors for ovarian cancer.

SECONDARY OUTCOMES:
Ovarian somatic mutations | 15 months
  To describe the presence of somatic mutations on ovarian tumor tissue, in patients with breast cancer arising during or after treatment with platinum-based chemotherapy or PARP-inhibitors for ovarian cancer.

CONTACTS AND LOCATIONS:
Locations (1):
- Fondazione Policlinico Universitario Agostino Gemelli IRCCS, Rome, RM, Italy

IPD SHARING:
Plan to Share IPD: No